CLINICAL TRIAL: NCT01651390
Title: BIOLUX RCT - Clinical Performance of the Pantera LUX Paclitaxel Releasing Balloon Versus the Drug Eluting Orsiro Hybrid Stent System in Patients With In-stent Restenosis - a Randomized Controlled Trial
Brief Title: Clinical Performance of the Pantera Lux Balloon Versus the Orsiro Stent in Patients With In-stent Restenosis.
Acronym: BIOLUX-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1105
Record Dates: First submitted 2012-07-24; First posted 2012-07-27 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Coronary Artery Disease; Coronary Restenosis
Keywords: Restenosis; Drug coated balloon; Drug eluting stent; Paclitaxel; Sirolimus
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug coated balloon (Experimental): Percutaneous coronary intervention with the Pantera Lux drug coated balloon.
  Interventions: Device: Percutaneous coronary intervention
- Drug eluting stent (Active Comparator): Percutaneous coronary intervention with the Orsiro drug eluting stent.
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — Up to 140 patients meeting the inclusion criteria and none of the exclusion criteria are randomly selected and stratified according to diabetic status at screening are treated with the Pantera Lux drug coated balloon.
  Other Names: Pantera Lux drug coated balloon; Paclitaxel; BTHC (Butyryltri-n-hexyl Citrate)
  Arms: Drug coated balloon
Device: Percutaneous coronary intervention — Up to 70 patients meeting the inclusion criteria and none of the exclusion criteria are randomly selected and stratified according to diabetic status at screening are treated with the Orsiro drug eluting stent.
  Other Names: Orsiro drug eluting stent; Orsiro hybrid drug eluting stent system; Sirolimus eluting stent
  Arms: Drug eluting stent

SUMMARY:
To determine in a randomized controlled trial (RCT) whether percutaneous coronary intervention - in patients with in-stent restenosis in either bare metal stents or drug eluting stents - with the Pantera Lux balloon is angiographically non-inferior to percutaneous intervention with the Orsiro stent 6 months post-procedure.

DETAILED DESCRIPTION:
This clinical investigation is an international, multi-center, randomized controlled trial with angiographic follow up at 6 months. Clinical follow ups will take place at 6, 12 and 18 months.

Up to 210 subjects will be block randomized 2:1 to receive the Pantera Lux balloon or the Orsiro stent and will be stratified according to diabetic status at screening.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided a written informed consent
2. Subject ≥ 18 years
3. Clinical evidence of ischemic heart disease and/or a positive functional study, stable or unstable angina pectoris or documented silent ischemia
4. Subject eligible for percutaneous coronary intervention
5. Subject acceptable candidate for coronary artery bypass surgery
6. Subject with an in-stent restenotic lesion* in either a bare metal stent or drug eluting stents (Mehran class I, II, III, IV - Mehran et al. Circulation 199; 100: 1872-1878). *Target lesion
7. Subjects with a maximum of 2 target lesions. In case of 2 target lesions, both lesions must be either in bare metal stents or drug eluting stents, and must treated during the same session with the same type of device as per randomization outcome, e.g. drug eluting stent.
8. Target reference vessel diameter (visual estimation): ≥ 2.0 and ≤ 4.0 mm
9. Target lesion length (visual estimation): ≥ 6.0 and ≤ 28.0 mm
10. Target lesion stenosis (visual estimation): > 50 % and ≤ 100 %
11. Target lesion in a native coronary artery

Exclusion Criteria:

1. Planned (staged) interventional treatment in the same vessel(s) as the target lesion(s) within 30 days pre- and/or post BIOLUX RCT index procedure.
2. Evidence of acute ST-segment-elevation myocardial infarction within 48 hours prior to index procedure according to the universal definition of myocardial infarction
3. Subjects with acute cardiac decompensation or acute cardiogenic shock
4. Subject with a life expectancy of less than 18 month
5. In the investigators opinion subject who will not be able to comply with the follow up requirements
6. Impaired renal function (excluded are subjects in need of dialysis or subjects with a creatinine level ≥ 221 µmol per liter (2.5 mg per deciliter) within 72 hours of the intended treatment)
7. Thrombus in the target vessel
8. Target lesion located in left main coronary artery
9. Documented left ventricular ejection fraction (LVEF) ≤ 30%
10. Known allergies to: acetylsalicylic acid, clopidogrel, prasugrel, ticagrelor, heparin, contrast medium, sirolimus or similar drugs (i.e., ABT 578, biolimus, tacrolimus); CoCr, PLLA, silicon carbide
11. Subject is receiving oral or intravenous immunosuppressive therapy (e.g., inhaled steroids are not excluded) or has known life-limiting immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus, but not including diabetes mellitus)
12. Subject currently enrolled in other investigational device or drug trial in which primary endpoint has not been reached
13. Pregnant and/or breast-feeding females or females who intend to become pregnant during the time of the study
14. Previously enrolled in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Late lumen loss (in-stent) | After 6 months.
  In-stent late lumen loss is defined as the difference between minimal luminal diameter after procedure and at 6 months, as evaluated by offline quantitative coronary angiography (QCA).
  In-stent:
  Pantera Lux balloon: In-stent is defined as from (proximal) shoulder to (distal) shoulder of the dilated balloon.
  Orsiro stent: In-stent is defined as from (proximal) edge to (distal) edge of the implanted Orsiro stent.

SECONDARY OUTCOMES:
Percent diameter stenosis in-stent and in-segment | After 6 months.
  Percent diameter stenosis is defined as the difference between reference vessel diameter and minimal lumen diameter divided by reference vessel diameter x100%. Angiographic parameters as evaluated by offline QCA.
  In-segment:
  Pantera Lux balloon: In-segment is defined as in-stent plus 5 mm distal and 5 mm proximal.
  Orsiro stent: In-segment is defined as in-stent plus 5 mm distal and 5 mm proximal.
Binary restenosis in-stent and in-segment | After 6 months.
  Binary restenosis is defined as ≥50% lumen diameter stenosis as evaluated by offline QCA.
Mean lumen diameter in-stent and in-segment | After 6 months.
  Mean minimum lumen diameter derived from two orthogonal views as evaluated by offline QCA.
Type of reoccurrence according to Mehran classification | After 6, 12 and 18 months.
  Type of reoccurrence according to Mehran classification (Mehran et al. Circulation 199; 100: 1872-1878) evaluated by offline QCA.
Target lesion failure (TLF) | After 6 and 18 months.
  TLF is defined as a composite of cardiac death, any target vessel myocardial infarction (MI), coronary artery bypass graft (CABG) and clinically driven target lesion revascularization (TLR).
Target vessel failure (TVF) | After 6, 12 and 18 months.
  TVF is defined as a composite of cardiac death, any target vessel myocardial infarction, coronary artery bypass graft and clinically driven target vessel revascularization (TVR).
Stent thrombosis | After 6, 12 and 18 months.
  According to Academic Research Consortium (ARC) definition (Cutlip et al. Circulation 2007; 115: 2344-2351).
Procedure success | During hospital stay or 7 days after procedure, whichever came first.
  Procedure success defined as achievement of a final diameter stenosis of <30% by QCA, using any percutaneous method, without the occurrence of death, MI, or repeat revascularization of the target lesion during the hospital stay or 7 days after procedure, whichever came first.
Device success | 1 day (During procedure)
  Successful delivery of the balloon or stent to the target lesion site in the coronary artery; and appropriate balloon inflation and deflation or stent deployment; and successful removal of the balloon or the delivery system.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph K Naber, MD, Principal Investigator — Contilia Heart- and Vascular Center, Elisabeth Krankenhaus, Klara-Kopp-Weg 1, 45138 Essen, Germany
Locations (14):
- Germany (13):
  - Universitäts-Herzzentrum Freiburg-Bad Krozingen, Bad Krozingen
  - Heart Center Segeberger Kliniken, Bad Segeberg
  - Charité - Universitätsmedizin Berlin, Charité Centrum 11 für Herz-, Kreislauf- und Gefäßmedizin, Berlin
  - Innere Medizin Kardiologie - Charité Centrum 11, Campus Benjamin Franklin, Berlin
  - Kardiologie - Angiologie - Pneumologie, Klinikum Coburg, Coburg
  - Contilia Heart- and Vascular Center, Elisabeth Krankenhaus, Essen
  - Medical Care Center Prof. Mathey, Prof. Schofer, Hamburg
  - Kardiologie /Intern. Intensivmedizin, Johannes Wesling Klinikum Minden, Minden
  - Klinikum Schwabing, Munich
  - LMU - Klinikum der Universität München, Munich
  - Klinikum Bogenhausen, Munich
  - Universitätsklinikum Münster, Klinik für Kardiologie, Münster
  - Innere Medizin III Kardiologie, Kliniken Villingen, Villingen-Schwenningen
- Cardiology, Pauls Stradins Clinical University Hospital, Riga, Latvia

REFERENCES:
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Background] Mehran R, Dangas G, Abizaid AS, Mintz GS, Lansky AJ, Satler LF, Pichard AD, Kent KM, Stone GW, Leon MB. Angiographic patterns of in-stent restenosis: classification and implications for long-term outcome. Circulation. 1999 Nov 2;100(18):1872-8. doi: 10.1161/01.cir.100.18.1872. PMID 10545431